CLINICAL TRIAL: NCT02316457
Title: First-in-human Clinical Study With RNA-Immunotherapy Combination of IVAC_W_bre1_uID and IVAC_M_uID for Individualized Tumor Therapy in Triple Negative Breast Cancer Patients
Brief Title: RNA-Immunotherapy of IVAC_W_bre1_uID and IVAC_M_uID
Acronym: TNBC-MERIT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Seventh Framework Programme (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BN_0002-01
Record Dates: First submitted 2014-11-21; First posted 2014-12-15 (Estimated); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer (Triple Negative Breast Cancer (TNBC))
Keywords: TNBC; Breast Cancer; Warehouse; Mutanome; RNA; Vaccine
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ARM1 IVAC_W_bre1_uID (Experimental): Patients enrolled in ARM1 will receive a treatment with four RNAs. This includes two to three variant RNAs selected from the WAREHOUSE plus p53 RNA. The selection process of RNAs from the warehouse is based on RT-PCR-based profiling of RNA extracted from patient tumor sample specimens, pre-defined cut-offs and algorithms to select the three relevant RNAs for a given patient.
  Interventions: Biological: IVAC_W_bre1_uID
- ARM2 IVAC_W_bre1_uID/IVAC_M_uID (Experimental): Patients enrolled in ARM2 will optionally receive the WAREHOUSE treatment as described above followed by the personalized IVAC® MUTANOME immunotherapy. The mutation selection process constitutes a multi-step process including identification of somatic mutations by NGS, mutation confirmation and prioritization, selection, and on demand manufacturing.
  Interventions: Biological: IVAC_W_bre1_uID/IVAC_M_uID
- ARM3 IVAC_W_bre1_uID + RBLTet.1 (Experimental): Patients enrolled in ARM3 will receive a treatment with four RNAs. This includes two to three variant RNAs selected from the WAREHOUSE plus p53 RNA. The selection process of RNAs from the warehouse is based on RT-PCR-based profiling of RNA extracted from patient tumor sample specimens, pre-defined cut-offs and algorithms to select the three relevant RNAs for a given patient. RBLTet.1 RNA will be added to each RNA applied.
  Interventions: Biological: IVAC_W_bre1_uID

INTERVENTIONS:
Biological: IVAC_W_bre1_uID — vaccination
  Arms: ARM1 IVAC_W_bre1_uID; ARM3 IVAC_W_bre1_uID + RBLTet.1
Biological: IVAC_W_bre1_uID/IVAC_M_uID — vaccination
  Arms: ARM2 IVAC_W_bre1_uID/IVAC_M_uID

SUMMARY:
The Mutanome Engineered RNA Immuno-Therapy (MERIT) study introduces a novel concept for Individualized Cancer Immunotherapy (IVAC®) to treat each patient with the relevant and immunogenic RNA vaccines for a given patient's tumor. The TNBC-MERIT trial uses two complementary strategies, the WAREHOUSE and the IVAC® MUTANOME concept, resulting in two custom-made IVAC® investigational medicinal products (IMPs) (IVAC_W_bre1_uID and IVAC_M_uID) for each individual patient.

DETAILED DESCRIPTION:
* The WAREHOUSE concept is based on RNA drug products shelved in a warehouse and targeting shared tumor-associated antigens (TAAs). The BioNTech Group (henceforward the "company") has identified a set of target antigens commonly expressed in TNBC. The selected breast cancer-associated antigens have been shown by immunogenicity testing to constitute suitable targets for immunotherapy and form the basis for the development of a novel RNA-based immunotherapy approach.
* The IVAC® MUTANOME concept is based on the identification of tumor-specific mutations by next-generation sequencing (NGS) and on-demand RNA manufacturing for use in single patients to target multiple neo-antigens derived from mutated epitopes. The novel therapeutic concept is supported by a series of research projects and high level publications that have led to a broad acceptance that mutation-specific T cells bear enormous potential to confer anti-tumoral activity in cancer patients.
* The TNBC-MERIT study will introduce the novel therapeutic concept for the individualized treatment of breast cancer that is based on (i) treatment with a patient-specific liposome complexed RNA tailored to the antigen-expression profile of any given patient's tumor (WAREHOUSE immunotherapy - IVAC_W_bre1_uID) and (ii) on treatment with de novo synthesized RNAs targeting up to 20 individual tumor mutations (IVAC® MUTANOME immunotherapy - IVAC_M_uID) following optional treatment with WAREHOUSE. The scientific rationale for the combination of the two IVAC® approaches is based on the assumption that immunotherapies that (1) acknowledge tumor heterogeneity on a single-patient level and (2) target the whole range of antigens selectively expressed on tumors ("cancer antigenome"), including immunogenic shared and unique antigens, bear the highest potential to constitute an effective treatment of tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive adenocarcinoma triple negative breast cancer (TNBC), pT1cN0M0 - anyTanyNM0 confirmed by physical examination or imaging
* Triple negative breast cancer is defined as:

  * HER2 negative
  * IHC 0-1+
  * IHC 2+ and FISH negative (ratio < 2.0 or < 4 gene copies / cell, as per new ASCO guideline)
  * ER and PR negative confirmed< 1%
* For patients with surgery of primary tumor followed by adjuvant chemotherapy, treatment with IVAC_W_bre1_uID will be initiated after completion of the adjuvant chemotherapy. The adjuvant chemotherapy should contain anthracyclines and taxanes - except for patients with contraindications for treatment with one or both substances.
* For patients with neoadjuvant chemotherapy according to local standard followed by surgery of primary tumor, treatment with IVAC_W_bre1_uID will be initiated after the surgery. The neoadjuvant chemotherapy should contain anthracyclines and taxanes - except for patients with contraindications for treatment with one or both substances.
* Patients with planned radiotherapy (as per local policy) are eligible and should be irradiated in parallel to the vaccination cycles
* Patients after completion of standard of care therapy e. g. surgery and/or chemotherapy and/or radiotherapy (as per local policy) are eligible at the discretion of the investigator after no clinical sings of recurrence and/or metastasis, if the treatment with IVAC_W_bre1_uID starts within one year after completion of the radiotherapy.
* Adequate organ function (hematopoietic, hepatic and renal function):

  * Hemoglobin ≥ 9 g/dl
  * ANC ≥ 1500/µl
  * Platelet count ≥ 100,000/mm³
  * ALT/AST <2 x ULN
  * Serum creatinine ≤ 1.5 ULN
* Expression of at least two tumor-specific antigens of the WAREHOUSE_bre1 confirmed by RT-qPCR on FFPE tumor tissue for ARM1 and ARM3
* Female patients, ≥ 18 years of age
* Written informed consent
* ECOG performance status (PS) 0-1
* Recovered pre-existing toxicities < grade 2 according to NCI CTCAE 4.03, except alopecia
* Negative pregnancy test (measured by β-HCG) for females of childbearing age
* Not pregnant or nursing

Exclusion Criteria:

* Patients with stage pT1a,bN0M0 and anyTanyNM1disease are excluded
* Patients with recurrence of breast cancer prior to the start of study treatment with IVAC_W_bre1_uID
* Any serious local infection (e. g. cellulitis, abscess) or systemic infection (e. g. pneumonia, septicemia, viral or fungal infection) which requires systemic treatment with antibiotics or corticoid therapy within two weeks prior to the first dose of study medication
* Previous splenectomy
* Concurrence of a second malignancy other than squamous or basal cell carcinoma or cervical carcinoma in situ within 5 years prior to the start of study treatment
* Known hypersensitivity to the active substance or to any of the excipients
* Prior solid organ transplantation or hematopoietic stem cell transplantation
* Positive test for acute Hepatitis A, acute or chronic active Hepatitis B or C infection
* Clinically relevant active autoimmune disease
* Systemic immune suppression:

  * HIV disease
  * Use of chronic oral or systemic steroid medication (topical or inhalational steroids are permitted)
  * Other clinically relevant systemic immune suppression
* Symptomatic congestive heart failure (NYHA 3 or 4)
* Unstable angina pectoris
* Adjuvant chemotherapy within 14 days before the first treatment of IVAC_W_bre1_uID
* Other major surgeries within 28 days before the first treatment
* Other investigational agents within 28 days or 5 half-lives depending on what gives the longer range before the first treatment
* Ongoing participation in another clinical study (except of Follow-Up observation)
* Fertile females who are unwilling to use a highly effective method of birth control (less than 1% per year, e.g. birth control pills, injections, patches, intrauterine device, or intrauterine hormone-releasing system) during study treatment and until End of Trial visit (EOT) at day 120
* Presence of a severe concurrent illness or another condition (e. g. psychological, family, sociological, or geographical circumstances) that does not permit adequate Follow-Up and compliance with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events as a Measure of Safety and Tolerability of IVAC_W_bre1_uID | day 120
  Assessment of AEs
Number of Adverse Events as a Measure of Safety and Tolerability of IVAC_W_bre1_uID plus IVAC_M_uID | up to day 246
  Assessment of AEs, End of treatment visit is depending on treatment schedule

SECONDARY OUTCOMES:
Change of induced T-cell responses for IVAC_W_bre_uID change from Visit 1 to V10 | up to 78 days
  Vaccine induced T-cell responses assessed by immuno assays in peripheral blood
Change of induced T-cell responses for IVAC_M_uID change from Visit 18 to Follow-up Visit | up to 78 days
  Vaccine induced T-cell responses assessed by immuno assays in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (4):
- Germany (3):
  - Johannes Gutenberg University, Mainz, RLP
  - National Center for Tumor Diseases (NCT), Heidelberg
  - Dr. Horst Schmidt-Kliniken Wiesbaden, Wiesbaden
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- See also: BioNTech SE — http://www.biontech.de